CLINICAL TRIAL: NCT02050594
Title: Ipilimumab 12-month Intensive Pharmacovigilance Protocol
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-366
Record Dates: First submitted 2014-01-14; First posted 2014-01-31 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Melanoma patients on Ipilimumab: All unresectable, recurrent or metastatic melanoma patients
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: Yervoy

SUMMARY:
The primary objective of the protocol is to identify and describe observed adverse events (AEs) while on treatment with Ipilimumab for advanced melanoma in Venezuela during the study period

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Age of 18 years or older on date of first dose of Ipilimumab
* Subjects who received at least 1 dose of Ipilimumab for the treatment of unresectable, recurrent or metastatic melanoma in Venezuela

Exclusion Criteria:

* Subjects who received Ipilimumab as part of a clinical trial
* Subjects who received Ipilimumab for any indication other than local approval (ie, unresectable or metastatic melanoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bristol Myers de Venezuela S.A.C. has in place a Customer Model registry, which tracks every Ipilimumab prescription in Venezuela. Therefore, any oncologist who treats a patient with Ipilimumab will be identified by BMS. Use of this registry will ensure all patients who are infused with Ipilimumab are included in this study
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Descriptive statistics of observed adverse events (AEs) while on treatment with Ipilimumab for advanced melanoma in Venezuela | Up to 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Caracas, Venezuela

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx